CLINICAL TRIAL: NCT05864040
Title: HYROS (HYbrid RObotic Surgery in Urology)
Brief Title: HYbrid RObotic Surgery in Urology
Acronym: HYROS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rob Surgical Systems S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PL-PR01-027
Record Dates: First submitted 2023-04-03; First posted 2023-05-18 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Nephrectomy
Keywords: Radical; Simple; Laparoscopy
MeSH Terms: conditions — Charcot-Marie-Tooth disease, Type 1C | interventions — Nephrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects to undergo laparoscopic radical/simple nephrectomy (Experimental): Adult subjects between 18 and 90 years old, that provided informed consent prior to any clinical investigation-related procedure, who have been scheduled for a laparoscopic radical/simple nephrectomy surgery and who are able and willing to comply with all study requirements to be evaluated for each study visit.
  Interventions: Device: Bitrack System-assisted laparoscopic radical/simple nephrectomy

INTERVENTIONS:
Device: Bitrack System-assisted laparoscopic radical/simple nephrectomy — Robot-Assisted Laparoscopic Transperitoneal Radical/Simple Nephrectomy is performed under general anesthesia. Using blunt dissection, the inferior pole of the kidney is lifted, and ureter and gonadal veins released from fat and connective tissue. The ureter is dissected caudally and sectioned after being sealed with a distal endoscopic clip. Dissection proceeds along the psoas muscle with anterior elevation of the ureter and lower renal pole towards the hilium. Main hilar are circumferentially dissected and sectioned and the kidney is entirely mobilized and released. Gerota´s capsule and suprarenal gland may be preserved if oncologically safe. Once the specimen is completely released, a laparoscopic bag is introduced by the assistant and the specimen entrapped. The robot is undocked, gas evacuated from the abdomen and specimen retrieved.

SUMMARY:
The HYbrid RObotic Surgery in urology (HYROS) study is an early feasibility clinical investigation of a new medical device under the commercial name of Bitrack System. Bitrack System is a surgical robot indicated to be used during urological surgical procedures. The Bitrack System also requires the specific single use of Electro-Surgical Endoscopic (ESE) instruments and Non-Electro Surgical Endoscopic (NESE) instruments.

The purpose of this clinical investigation is to evaluate the safety and feasibility of the Bitrack System and its corresponding ESE and NESE instruments in patients with the indication of a robot assisted laparoscopic radical/simple nephrectomy.

DETAILED DESCRIPTION:
The Bitrack System is a surgical robot indicated to be used during urological surgical procedures. This robot is intended to assist in the accurate control of endoscopic instruments and accessories for visualization and endoscopic manipulation.

Robotic Assisted Surgical (RAS) systems and equipment such as Bitrack System are intended for use in invasive surgical procedures, during which patients are potentially most vulnerable to physical harm. The Bitrack System comprises a console, a robotic unit, and embedded software.

The HYROS clinical investigation will be conducted as a single-center, early feasibility, and first-in-human (FIH) clinical investigation with a single arm, open-label, and non-randomized design, that will include 3 patients. This clinical investigation aims to evaluate the safety and performance of the Bitrack System in patients indicated with robotic-assisted laparoscopic Radical/simple nephrectomy surgery.

The planned visits for this clinical investigation are baseline (includes Screening, baseline visit, and Informed consent), procedure, discharge, 14-Days Follow-up visit, and 30-Days Follow-up visit (remote). The clinical investigation will include adult subjects (between 18 and 90 years old) who have been scheduled for laparoscopic radical/simple nephrectomy. The total duration of the clinical investigation is expected to be 4 months, consisting of approximately 3 months of enrollment plus 1 month of follow-up. The end of the clinical investigation will occur when the last visit of the last enrolled subject is completed.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects between 18 and 90 years old
* Subjects must provide written informed consent prior to any clinical investigation related procedure
* Subjects who have been scheduled for a laparoscopic radical/simple nephrectomy surgery
* Ability and willingness to comply with all study requirements to be evaluated for each study visit

Exclusion Criteria:

* Pregnant or breastfeeding women at the time of the surgery
* Inability to adhere to study-related procedures
* Subject has known allergy to some of the device components (i.e., stainless steel, etc.)
* Subjects who participate in another trial which may affect the outcome data on this study or the ability to complete the follow-up requirements
* Subjects not suitable to undergo MIS (Minimally Invasive Surgery) /MIRS (Minimally Invasive Robotic Surgery), according to medical criteria
* Subjects with life expectancy inferior to 3 months
* Subjects with a Body Mass Index (BMI) ≥ 40
* Subjects with severe cardiopulmonary or coronary artery disease, bleeding disorders or that have been submitted to multiple prior operations
* Subjects with abuses of active substances or with uncontrolled psychiatric disorders
* Subjects scheduled for surgeries intended to be in direct contact with the heart, the central circulatory system or the central nervous system
* Subjects with any contraindication for the use of the Bitrack System and the ESE/NESE instruments, as specified in the Instructions For Use

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lluis Peri Cusi, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy: Adult subjects between 18 and 90 years old, that provided informed consent prior to any clinical investigation-related procedure, who have been scheduled for a laparoscopic radical/simple nephrectomy surgery and who are able and willing to comply with all study requirements to be evaluated for each study visit. Robot-Assisted Laparoscopic Transperitoneal Radical/Simple Nephrectomy is performed under general anesthesia.
Period: Overall Study
Arm/Group | Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy
Number analyzed (Participants) | 3
Age, Customized [Number; unit: years] — Age at enrolment
  years
    Subject 01 | 53
    Subject 02 | 49
    Subject 03 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Safety of the Bitrack System
Description: Evaluation of the safety of the Bitrack System by measuring the occurrence of Procedure-Related Adverse Events (PRAEs) and Serious Adverse Events (SAEs) during the procedure and through the 30 days post-procedure period of enrolled patients indicated for robot assisted laparoscopic radical/simple nephrectomy. PRAEs are defined as any AE related to the investigational procedure.
Time Frame: 30 days post-procedure
Measure: Number; unit: adverse events
Arm/Group | Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy
Number analyzed (Participants) | 3
adverse events
  PRAEs through 30 days | 0
  SAEs through 30 days | 0

2. Primary Outcome: Performance of the Bitrack System
Description: Evaluation of the performance of the investigational device by means of its ability to access and reach the target zone, perform all relevant surgical tasks and to be withdrawn efficiently without conversion to minimally invasive surgery (MIS) or open surgery. The performance of the Bitrack System and the ESE/NESE instruments is analyzed through the conversion rate to conventional laparoscopy/open surgery.
Time Frame: During the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy
Number analyzed (Participants) | 3
Participants
  Surgery successfully completed with the Bitrack System | 3
  Conversion to open surgery | 0
  Conversion to laparoscopic surgery | 0

3. Secondary Outcome: Number of Participants With Adverse Events
Description: All AE(s) events during the procedure and through the 14 and 30 days post-procedure were also assessed, including the assessment of the relationship with the investigational device and/or procedure by the principal investigator.
Time Frame: Procedure, discharge (up to one week post-procedure), 14 days and 30 days follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy
Number analyzed (Participants) | 3
Participants
  Adverse Event (AE) reported | 0
  Mild AE | 0
  Moderate AE | 0
  Severe AE | 0
  Device-related AE | 0
  Procedure-related AE | 0
  Other AE according to relationship to the study | 0

4. Secondary Outcome: Number of Participants With Absence of Tissue Damage
Description: Individual safety is defined as absence of unwanted injure of any tissue for each instrument.
Time Frame: During the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy
Number analyzed (Participants) | 3
Participants | 3

5. Secondary Outcome: Individual Performance of Surgical Instruments
Description: Individual performance is assessed by the Visual Analogue Scale (ranging from 0 to 10) following the subjective surgeon's opinion for each instrument surgical function, being 0 a non-functional tool and 10 an instrument that works exactly equivalent to the surgeon/s hands.
Time Frame: During the procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy
Number analyzed (Participants) | 3
score on a scale | 7.33 (1.23)

6. Secondary Outcome: Blood Loss
Description: Blood Loss defined as estimated mL of blood loss
Time Frame: During the procedure
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy
Number analyzed (Participants) | 3
mL | 183.33 (125.83)

7. Secondary Outcome: Transfusion Rates
Description: Transfusion rate as the number of participants that required blood transfusion
Time Frame: During the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy
Number analyzed (Participants) | 3
Participants | 0

8. Secondary Outcome: Number of Participants That Require Hemostatic Agents.
Description: Number of participants that require the use of hemostatic agents.
Time Frame: During the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy
Number analyzed (Participants) | 3
Participants | 0

9. Secondary Outcome: Operative Time Procedure
Description: Operative Time Procedure (or Surgical Procedure Time) includes the time spend to perform the set of all the different tasks completed during the surgical procedure. It is defined from first ESE/NESE instruments docking to the conversion to gestural mode for their final withdrawal.
Time Frame: During the entire surgical procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy
Number analyzed (Participants) | 3
minutes | 123.6 (40.79)

10. Secondary Outcome: Post-operative Pain
Description: Evaluation of the post-operative pain in patients through the Cumulative Analgesic Consumption Score (CACS) during the first week (7days) post-procedure.
  To calculate the CACS score, information on the number of single analgesic doses (n) and their classification on the WHO pain relief ladder was collected. The WHO pain relief ladder ranges from I to III:
  * step I (nonopioids): acetaminophen, ibuprofen or metamizole;
  * step II (opioids for mild to moderate pain): tramadol, tilidine/naloxone;
  * step III (opioids for moderate to severe pain): piritramide, pethidine, oxycodone or morphine.
  The Cumulative Analgesic Consumption Score (CACS) is calculated by adding all (n), multiplied by the level of the WHO pain relief ladder.
  Since the lenght of stay was shorter (2-3 days), it was not possible to collect the analgesic consumption up to 7 days after patient hospital discharge.
Time Frame: Day 1 and Day 2 post-procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects to Undergo Laparoscopic Radical/Simple Nephrectomy
Number analyzed (Participants) | 3
units on a scale
  Day 1 | 4.67 (3.78)
  Day 2 | 3.33 (2.31)

11. Secondary Outcome: Length of Stay (LoS) in Hospital
Description: Assessment of the duration of subject's hospitalization as the Length of Stay (LoS) in hospital calculated from day of admission to day of discharge.
Time Frame: Discharge (up to one week post-procedure)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy
Number analyzed (Participants) | 3
days | 2.33 (0.58)

12. Secondary Outcome: Patient Pain Assessment
Description: Patient pain assessment via Visual Analog Score (VAS) for pain on a scale from 0 ('no pain') to 10 ('pain as bad as it could possibly be').
Time Frame: Discharge (up to one week post-procedure), 14- and 30-days post-procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy
Number analyzed (Participants) | 3
score on a scale
  Discharge | 4 (1.73)
  Day 14 | 1 (0)
  Day 30 | 0.67 (1.15)

13. Secondary Outcome: Post-procedure Complication Rates - Comprehensive Complication Index (CCI)
Description: Post-procedure complication rates assessment by measuring the Comprehensive Complication Index (CCI) on a scale from 0 (no complications) to 100 (death).
Time Frame: Discharge (up to one week post-procedure),14 and 30 days follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy
Number analyzed (Participants) | 3
score on a scale
  Discharge | 0 (0)
  Day 14 | 0 (0)
  Day 30 | 0 (0)

14. Secondary Outcome: Post-procedure Complication Rates - Clavien-Dindo Classification
Description: Post-procedure complication rates assessment by the Clavien-Dindo classification, which consists of 7 grades (I, II, IIIa, IIIb, Iva, Ivb and V), the first one (I) indicating any deviation from the normal postoperative course and the highest (V) corresponding to death.
Time Frame: Discharge (up to one week post-procedure),14 and 30 days follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy
Number analyzed (Participants) | 3
Participants
  Subject 01 | NA — No post-procedure complications were reported, and therefore classification was not applicable
  Subject 02 | NA — No post-procedure complications were reported, and therefore classification was not applicable
  Subject 03 | NA — No post-procedure complications were reported, and therefore classification was not applicable

ADVERSE EVENTS:
Time Frame: From baseline to 30-days post-procedure.
Description: All Adverse Events during the procedure and through the 14- and 30-days post-procedure were assessed. The relationship with the investigational device and/or procedure was examined by the Principal Investigator and reported to the Sponsor.
Arm/Group | Bitrack System-assisted Laparoscopic Radical/Simple Nephrectomy
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT05864040/Prot_000.pdf